CLINICAL TRIAL: NCT05636865
Title: Descriptive Study of the Incidence and Outcome of PAS in Two Large Referral Hospitals in Egypt , Kasr Alainy Hospital , Cairo University , and Banisuef Specialized Hospital in Last 6 Years
Brief Title: Descriptive Study of the Incidence and Outcome of PAS in Two Large Referral Hospitals in Egypt
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rihab Hagag Sayed, resident doctor , principle investigator, Cairo University
Other Study IDs: MS-26-2022
Record Dates: First submitted 2022-11-13; First posted 2022-12-05 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-11

CONDITIONS: Placenta Accreta
Keywords: PAS
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
placenta accreta spectrum incidence and outcome

DETAILED DESCRIPTION:
placenta accreta spectrum ( PAS ) one of the most serious condition in obstetrics nowadays so the investigators measure the incidence by this study

ELIGIBILITY:
Inclusion Criteria:

* gestational age above 28 weeks

Exclusion Criteria:

* age less than 18

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes
Study Population: pregnant woman above 28 weeks
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2022-07-30 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
number of diagnosed pregnant women with placenta accreta spectrum | in last 6 years
  pregnant women with gestitional age above 18 week , with confirmed diagnosis with PAS with U/S

SECONDARY OUTCOMES:
incidence of hystrectomy | in last 6 years
  hystrectomy VS conservative management

CONTACTS AND LOCATIONS:
Overall Officials: rihab hagag, resident, Principal Investigator — kasr alainy
Locations (1):
- Kasr Alainy , Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
incidence of PAS